CLINICAL TRIAL: NCT00328614
Title: A Phase I Pilot Study of Samarium-153 Combined With Neoadjuvant Hormonal Therapy and Radiation Therapy in Men With Locally Advanced Prostate Cancer
Brief Title: Samarium-153 With Neoadjuvant Hormonal and Radiation Therapy for Locally Advanced Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Cytogen Corporation (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02C.172; 2001-114 (Other: CCRRC); JT 1013 (Other: JeffTrial Number)
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Locally advanced prostate cancer; positive lymph nodes
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Samarium-153; samarium Sm-153 lexidronam; 3,5-tetrahydroaldosterone sulfate; bicalutamide; Goserelin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Samarium-153 (0.25 mCi/kg) (Experimental): Cohort 1: Patients receive 0.25 mCi/kg of Samarium-153, hormonal therapy, and radiation therapy
  Interventions: Drug: Samarium-153; Drug: Total Androgen Suppression (TAS) with Bicalutamide; Drug: Total androgen suppression (TAS) with Goserelin Acetate; Device: Radiation Therapy
- Samarium-153 (0.5 mCi/kg) (Experimental): Cohort 2: Patients receive 0.5 mCi/kg of Samarium-153, hormonal therapy, and radiation therapy
  Interventions: Drug: Samarium-153; Drug: Total Androgen Suppression (TAS) with Bicalutamide; Drug: Total androgen suppression (TAS) with Goserelin Acetate; Device: Radiation Therapy
- Samarium-153 (0.75 mCi/kg) (Experimental): Cohort 3: Patients receive 0.75 mCi/kg of Samarium-153, hormonal therapy, and radiation therapy
  Interventions: Drug: Samarium-153; Drug: Total Androgen Suppression (TAS) with Bicalutamide; Drug: Total androgen suppression (TAS) with Goserelin Acetate; Device: Radiation Therapy
- Samarium-153 (1.0 mCi/kg) (Experimental): Cohort 4: Patients receive 1.0 mCi/kg of Samarium-153, hormonal therapy, and radiation therapy
  Interventions: Drug: Samarium-153; Drug: Total Androgen Suppression (TAS) with Bicalutamide; Drug: Total androgen suppression (TAS) with Goserelin Acetate; Device: Radiation Therapy
- Samarium-153 (1.5 mCi/kg) (Experimental): Cohort 5: Patients receive 1.5 mCi/kg of Samarium-153, hormonal therapy, and radiation therapy
  Interventions: Drug: Samarium-153; Drug: Total Androgen Suppression (TAS) with Bicalutamide; Drug: Total androgen suppression (TAS) with Goserelin Acetate; Device: Radiation Therapy
- Samarium-153 (2.0 mCi/kg) (Experimental): Cohort 6: Patients receive 2.0 mCi/kg of Samarium-153, hormonal therapy, and radiation therapy
  Interventions: Drug: Samarium-153; Drug: Total Androgen Suppression (TAS) with Bicalutamide; Drug: Total androgen suppression (TAS) with Goserelin Acetate; Device: Radiation Therapy

INTERVENTIONS:
Drug: Samarium-153 — Samarium-153 will be administered as a single dose after one month of hormonal therapy. The dose level of Samarium-153 may change to determine maximum tolerated dose (MTD).
  Other Names: Samarium-153-ethylene diamine tetramethylene phosphonate; Samarium (153Sm) lexidronam; Quadramet
Drug: Total Androgen Suppression (TAS) with Bicalutamide — Patients will receive 5 months of total androgen suppression (TAS) consisting of Zoladex and Casodex. Total androgen suppression will begin 3 months prior to initiation of irradiation.
  Other Names: Casodex
Drug: Total androgen suppression (TAS) with Goserelin Acetate — Patients will receive 5 months of total androgen suppression (TAS) consisting of Zoladex and Casodex. Total androgen suppression will begin 3 months prior to initiation of irradiation.
  Other Names: Zoladex
Device: Radiation Therapy — Radiation therapy will begin 3 months following the initiation of hormone administration. Daily tumor doses will be given 5 days per week for 7-8 weeks.
  Other Names: XRT; Radiotherapy

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of Samarium-153 when given in combination with hormonal and external beam radiation therapy in men with high risk prostate cancer.

DETAILED DESCRIPTION:
The likelihood of prostate cancer cells metastasizing to bone has an early and important influence on the natural history of prostate cancer. Bone-targeted therapy, when given sequentially with hormonal therapy (androgen suppression) and radiation therapy, prolongs the progression of the disease in clinically non-metastatic prostate cancer patients.

The use of Samarium-153 EDTMP in conjunction with hormonal therapy and external beam radiation therapy has never been previously evaluated in high risk clinically localized prostate cancer. Many patients with high-risk prostate cancer develop progressive disease within 2 years of therapy indicating that subclinical metastatic disease may be present at the time of initial diagnosis. In these high-risk patients, there may be a therapeutic benefit of combining hormonal therapy with external beam radiation therapy and Samarium-153 EDTMP to treat localized and subclinical bony disease, respectively.

ELIGIBILITY:
Inclusion Criteria:

* PSA 20-150 and Gleason score greater than or equal to 7 or clinical stage greater than or equal to T2, Gleason greater than or equal to 8, PSA less than or equal to 150
* Pathologically positive lymph nodes
* Pretreatment must be prior to study entry and prior to any hormonal therapy
* Zubrod 0-1
* Adequate hematologic function

Exclusion Criteria:

* Patients with PSA equal to or greater than 150
* Neuroendocrine features on histologic examination
* Radiologic evidence of metastatic disease
* Previous malignancy within last 5 years
* Prior pelvic radiation therapy or orchiectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-03; Primary Completion 2009-02 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Trabulsi, MD, Principal Investigator — Thomas Jefferson University; Richard Valicenti, MD, MA, Study Chair — UC Davis School of Medicine
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Samarium-153 (0.25 mCi/kg) | Samarium-153 (0.5 mCi/kg) | Samarium-153 (0.75 mCi/kg) | Samarium-153 (1.0 mCi/kg) | Samarium-153 (1.5 mCi/kg) | Samarium-153 (2.0 mCi/kg)
Started | 4 | 4 | 6 | 6 | 6 | 6
Completed | 4 | 4 | 6 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Samarium-153 (0.25 mCi/kg) | Samarium-153 (0.5 mCi/kg) | Samarium-153 (0.75 mCi/kg) | Samarium-153 (1.0 mCi/kg) | Samarium-153 (1.5 mCi/kg) | Samarium-153 (2.0 mCi/kg) | Total
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 6 | 6 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 3 | 1 | 3 | 2 | 10
  >=65 years | 4 | 3 | 3 | 5 | 3 | 4 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.97 (1.37) | 65.10 (9.78) | 65.58 (10.00) | 69.46 (8.04) | 68.00 (13.13) | 66.19 (8.02) | 66.99 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 4 | 6 | 6 | 6 | 6 | 32
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 6 | 6 | 6 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Samarium-153
Description: To determine the maximum tolerated dose (MTD) of Samarium as adjuvant to combined hormonal therapy (HT) and external beam radiation therapy (RT).
  Dose levels:
  Dose I: 0.25 mCi/kg IV Dose II: 0.5 mCi/kg IV Dose III: 0.75 mCi/kg IV Dose IV: 1.0 mCi/kg IV Dose V: 1.5 mCi/kg IV Dose VI: 2.0 mCi/kg IV
  Dose-limiting toxicity will be defined as Grade 3 hematologic toxicity per NCI Common Toxicity Criteria. The maximally tolerated dose (MTD) will then be the last dose studied or the previous dose, based on clinical judgment of the degree of toxicity seen at the last dose.
Time Frame: 5 months (1 month HT, administration of drug, 4 months HT and RT)
Measure: Number; unit: mCi/kg
Groups:
- Samarium-153: Cohort 1: Patients receive 0.25 mCi/kg of Samarium-153, hormonal therapy, and radiation therapy
Arm/Group | Samarium-153
Number analyzed (Participants) | 29
mCi/kg | 2.0

ADVERSE EVENTS:
Arm/Group | Samarium-153 (0.25 mCi/kg) | Samarium-153 (0.5 mCi/kg) | Samarium-153 (0.75 mCi/kg) | Samarium-153 (1.0 mCi/kg) | Samarium-153 (1.5 mCi/kg) | Samarium-153 (2.0 mCi/kg)
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4 | 1/6 | 2/5 | 3/5 | 5/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/6 | 0/5 | 0/5 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Samarium-153 (0.25 mCi/kg) (N=4) | Samarium-153 (0.5 mCi/kg) (N=4) | Samarium-153 (0.75 mCi/kg) (N=6) | Samarium-153 (1.0 mCi/kg) (N=5) | Samarium-153 (1.5 mCi/kg) (N=5) | Samarium-153 (2.0 mCi/kg) (N=6)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 5 (5)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Blood/bone marrow (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Platelet count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 5 (5)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine color changed (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain and cramping (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flashes/flushes (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes